CLINICAL TRIAL: NCT06602921
Title: Does Dietary Nitrate Supplementation Attenuate the Cardiovascular Strain Elicited by Caffeine and Cold Exposure in Healthy Individuals?
Brief Title: The Effects of Nitrate, Caffeine, and Cold Exposure on Cardiovascular Function.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loughborough University (Other)
Collaborators: Biogen Extracts Pvt Ltd (Unknown)
Responsible Party: Principal Investigator, Stephen Bailey, Principal Investigator, Loughborough University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: LoughboroughUAM
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2024-08

CONDITIONS: Nitrate; Caffeine; Cold Exposure
Keywords: Cardiovascular Function; Flow mediated dilation
MeSH Terms: interventions — Caffeine

STUDY DESIGN:
Intervention Model Description: 24 participants will complete 4 experimental conditions in a randomized order.
Who Masked: Participant, Investigator
Masking Description: Double-blinded using supplement placebos.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Nitrate, caffeine, and cold pressor test (CPT) (Experimental): All outcome variables will be measured for 24 participants in a trial where they receive 400 mg nitrate in the form of beetroot extract, 6 mg/kg caffeine powder, and undergo a 3 min cold pressor test.
  Interventions: Dietary Supplement: TruBeet inorganic beetroot juice; Dietary Supplement: Caffeine; Other: Cold pressor test
- Nitrate, placebo caffeine, and CPT (Placebo Comparator): All outcome variables will be measured for 24 participants in a trial where they receive 400 mg nitrate in the form of beetroot extract, 6 mg/kg cornflour (caffeine placebo), and undergo a 3 min cold pressor test.
  Interventions: Dietary Supplement: TruBeet inorganic beetroot juice; Other: Cold pressor test
- Placebo nitrate, caffeine, and CPT (Placebo Comparator): All outcome variables will be measured for 24 participants in a trial where they receive nitrate-depleted beetroot extract (placebo), 6 mg/kg caffeine powder, and undergo a 3 min cold pressor test.
  Interventions: Dietary Supplement: Caffeine; Other: Cold pressor test
- Placebo nitrate, placebo caffeine, and CPT (Placebo Comparator): All outcome variables will be measured for 24 participants in a trial where they receive nitrate-depleted beetroot extract (placebo), 6 mg/kg cornflour (caffeine placebo), and undergo a 3 min cold pressor test.
  Interventions: Other: Cold pressor test

INTERVENTIONS:
Dietary Supplement: TruBeet inorganic beetroot juice — 400 mg nitrate-rich beetroot powder, mixed with 300 mL water.
  Arms: Nitrate, caffeine, and cold pressor test (CPT); Nitrate, placebo caffeine, and CPT
Dietary Supplement: Caffeine — 6 mg/kg caffeine powder in capsule form.
  Arms: Nitrate, caffeine, and cold pressor test (CPT); Placebo nitrate, caffeine, and CPT
Other: Cold pressor test — 3 min cold pressor test using the left foot in cold water (0-2 degree).

SUMMARY:
Dietary inorganic nitrate supplementation may have positive implications on cardiovascular function. The aim of this project is to determine if nitrate supplementation can attenuate the effects that caffeine and cold exposure have on the cardiovascular system.

DETAILED DESCRIPTION:
Acute caffeine consumption and cold exposure elicit negative effects on the cardiovascular system. Humans are regularly exposed to such conditions of increased cardiovascular strain, which may lead to elevated chronic cardiovascular risk. On the other hand, dietary inorganic nitrate supplementation is well established to improve cardiovascular function in healthy individuals. Thus, acute nitrate supplementation may compensate for the negative effects that caffeine and the cold place on the cardiovascular system. These effects will be measured using peripheral blood pressure, pulse wave analysis, heart rate variability, forearm blood flow, flow mediated dilation, and blood and saliva markers.

ELIGIBILITY:
Inclusion Criteria:

* Blood pressure < 130 mmHg systolic and < 85 mmHg diastolic. BMI between 18.5 and 29.9 kg/m2. Females must be naturally menstruating (regular length cycle and menses) or using a form of combined hormonal contraception (for at least 6 months).

Exclusion Criteria:

* Existing cardiovascular or metabolic conditions. Experience any adverse reactions to experimental procedures or supplements. Allergies to supplements or breakfast items. Involved in any other studies. Blood pressure > 130 mmHg systolic and > 85 mmHg diastolic.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-12-05 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Brachial blood pressure | Mean of 5 readings taken pre-supplementation (0 hours) and post-supplementation (2.5 hours). 1 reading was taken pre- cold pressor test (3.5 hours). All measures were recorded on every experimental trial (4 trials with at least 48 h washout between).
  Brachial blood pressure was collected using an automatic sphygmomanometer.
Flow mediated dilation | Measured pre-supplementation (at 0 hours) and post-supplementation (at 2.5 hours) for every experimental trial (4 trials with at least 48 h washout between).
  Baseline diameter, peak diameter, change in diameter, and shear stimulus following flow mediated dilation procedure of the brachial artery with post-occlusion reactive hyperaemia.
Central blood pressure and pulse wave variables | Collected pre-supplementation (0 hours), post-supplementation (2.5 hours), and during the cold pressor test (3.5 h) for 4 experimental trials (4 trials with at least 48 hours washout in between).
  Mean of 2-3 readings for aortic systolic BP, aortic diastolic BP, HR, Augmentation index, augmentation index corrected to HR of 75 bpm, pulse pressure, and augmentation pressure.

SECONDARY OUTCOMES:
Forearm blood flow | Measured pre-supplementation (at 0 hours) and post-supplementation (at 2.5 hours) for every experimental trial (4 trials with at least 48 h washout between).
  Forearm blood flow pre- and post-PORH (post occlusion reactive hyperaemia) via strain gauge plethysmography.
Salivary nitrate and nitrite | Measured pre-supplementation (at 0 hours) and post-supplementation (at 2.5 hours) for every experimental trial (4 trials with at least 48 h washout between).
  Salivary concentration of nitrate and nitrite
Heart rate variability | Collected pre-supplementation (0 hours), post-supplementation (2.5 hours), and during the cold pressor test (3.5 h) for 4 experimental trials (4 trials with at least 48 hours washout in between).
  Time and frequency domains for heart rate variability collected for 3-5min.
NIBP continuous blood pressure | Collected pre-supplementation (0 hours), post-supplementation (2.5 hours), and during the cold pressor test (3.5 h) for 4 experimental trials (4 trials with at least 48 hours washout in between).
  SBP, DBP, MAP, HR collected continuously for 3-5 min.
Whole blood RSNO | Collected pre-supplementation (0 hours), post-supplementation (2.5 hours), and immediately post- cold pressor test (3.5 h) for 4 experimental trials (4 trials with at least 48 hours washout in between).
  S--nitrosothiols concentration from treated whole blood (NEM, EDTA, potassium ferricyanide).
Plasma nitrate, nitrite, cGMP | Collected pre-supplementation (0 hours), post-supplementation (2.5 hours), and immediately post- cold pressor test (3.5 h) for 4 experimental trials (4 trials with at least 48 hours washout in between)
  Plasma concentrations of nitrate, nitrite, and cGMP.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Bailey, Principal Investigator — Loughborough University
Locations (1):
- Loughborough University, Loughborough, United Kingdom

IPD SHARING:
Plan to Share IPD: No